CLINICAL TRIAL: NCT02080650
Title: Characterization of Circulating Tumor Cells Captured by c-MET (CTC-MET)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: Prostate Cancer Foundation (Other); Janssen Diagnostics, LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: Pro00052149
Record Dates: First submitted 2014-03-03; First posted 2014-03-06 (Estimated); Last update posted 2017-08-01 (Actual); Status verified 2017-07

CONDITIONS: Prostate Cancer; Renal Cell Carcinoma; Bladder Cancer; Colorectal Cancer; Gastric Cancer; Pancreatic Cancer; Non-small Cell Lung Cancer; Advanced MET Amplified Solid Tumor
MeSH Terms: conditions — Prostatic Neoplasms; Carcinoma, Renal Cell; Urinary Bladder Neoplasms; Colorectal Neoplasms; Stomach Neoplasms; Pancreatic Neoplasms; Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (8):
- Prostate cancer (Other): Mesenchymal-marker based ferrofluid (c-MET)
  Interventions: Device: Mesenchymal-marker based ferrofluid (c-MET); Device: Epithelial cell adhesion molecule (EpCAM) ferrofluid
- Renal cell carcinoma (Other): Mesenchymal-marker based ferrofluid (c-MET)
  Interventions: Device: Mesenchymal-marker based ferrofluid (c-MET); Device: Epithelial cell adhesion molecule (EpCAM) ferrofluid
- Bladder cancer (Other): Mesenchymal-marker based ferrofluid (c-MET)
  Interventions: Device: Mesenchymal-marker based ferrofluid (c-MET); Device: Epithelial cell adhesion molecule (EpCAM) ferrofluid
- Gastric cancer (Other): Mesenchymal-marker based ferrofluid (c-MET)
  Interventions: Device: Mesenchymal-marker based ferrofluid (c-MET); Device: Epithelial cell adhesion molecule (EpCAM) ferrofluid
- Colorectal cancer (Other): Mesenchymal-marker based ferrofluid (c-MET)
  Interventions: Device: Mesenchymal-marker based ferrofluid (c-MET); Device: Epithelial cell adhesion molecule (EpCAM) ferrofluid
- Pancreatic cancer (Other): Mesenchymal-marker based ferrofluid (c-MET)
  Interventions: Device: Mesenchymal-marker based ferrofluid (c-MET); Device: Epithelial cell adhesion molecule (EpCAM) ferrofluid
- Non-small cell lung cancer (Other): Mesenchymal-marker based ferrofluid (c-MET)
  Interventions: Device: Mesenchymal-marker based ferrofluid (c-MET); Device: Epithelial cell adhesion molecule (EpCAM) ferrofluid
- Advanced MET amplified solid tumor (Other): Mesenchymal-marker based ferrofluid (c-MET)
  Interventions: Device: Mesenchymal-marker based ferrofluid (c-MET); Device: Epithelial cell adhesion molecule (EpCAM) ferrofluid

INTERVENTIONS:
Device: Mesenchymal-marker based ferrofluid (c-MET)
Device: Epithelial cell adhesion molecule (EpCAM) ferrofluid

SUMMARY:
This pilot study will aim to determine whether circulating tumor cells (CTCs) can be captured using the novel cMET based ferrofluid. The primary objective of this pilot study will be to describe the numbers of c-MET expressing cells that can be detected by the c-MET CTC capture technique. These data will be separated by disease site. The investigator will also describe the detection rates of both the c-MET CTC capture and the EpCAM CTC capture techniques in each patient, also separated by disease site.

ELIGIBILITY:
Inclusion Criteria:

Prostate cancer patients will be eligible for inclusion in this study only if all of the following criteria apply:

1. Histologically confirmed diagnosis of adenocarcinoma of the prostate. Small cell or neuroendocrine tumors of the prostate are also permitted.
2. Clinical or radiographic evidence of metastatic disease.
3. Castrate levels of testosterone (<50 ng/dl)
4. Enrollment prior to the initiation of a new systemic therapy.
5. Evidence of disease progression on or following most recent therapy as evidenced by either of the following:

   * Two consecutive PSA levels greater than the PSA nadir achieved on ADT and most recent therapy, separated by greater than one week
   * Radiographic evidence of disease progression as defined by new bone scan lesions or growth of soft tissue/visceral metastases >1 cm in diameter (2 cm for lymph nodes).
   * Clinical progression of disease with cutaneous lesions or palpable lesions in absence of radiographic progression
6. Age > 18 years.
7. Ability to understand and the willingness to sign a written informed consent document.

Renal cell carcinoma patients will be eligible for inclusion in this study only if all of the following inclusion criteria apply:

1. Histologically confirmed diagnosis of invasive renal cell carcinoma (all histologies)
2. Clinical or radiographic evidence of metastatic disease.
3. Evidence of disease progression on the current or following the most recent therapy, as defined by one of the following:

   * A new soft tissue/visceral/lymph node/bone metastatic lesion
   * Growth of existing soft tissue/visceral/lymph node/bone metastases as determined by the investigator
   * Clinical progression of disease with cutaneous lesions or palpable lesions in absence of radiographic progression
4. For clear cell carcinoma, refractory to treatment with VEGF inhibitors as defined by progression on VEGF therapy within 1 year of starting VEGF therapy. For non-clear cell histologies, any line of systemic therapy.
5. Enrollment prior to the initiation of a new systemic therapy.
6. Age > 18 years.
7. Ability to understand and the willingness to sign a written informed consent document.

Bladder cancer patients will be eligible for inclusion in this study only if all of the following inclusion criteria apply:

1. Histologically confirmed diagnosis of invasive bladder transitional cell carcinoma, adenocarcinoma, squamous cell carcinoma, or small cell carcinoma.
2. Metastatic disease with either bone or visceral metastatic lesions, or clinically symptomatic with metastatic disease.
3. Progression of disease on or following the most recent treatment as evidenced by one of the following:

   * A new soft tissue/visceral/lymph node/bone metastatic lesion
   * Growth of existing soft tissue/visceral/lymph node/bone metastases as determined by the investigator.
   * Clinical progression of disease with cutaneous lesions, palpable lesions, pleural effusions, or ascites in absence of radiographic progression
4. Enrollment prior to the initiation of a new systemic therapy.
5. Age > 18 years.
6. Ability to understand and the willingness to sign a written informed consent document.

Gastric cancer (including gastroesophageal junction) patients will be eligible for inclusion in this study only if all of the following inclusion criteria apply:

1. Histologically confirmed diagnosis of invasive gastric or distal esophageal adenocarcinoma.
2. Clinical or radiographic evidence of metastatic disease.
3. Evidence of disease progression on or following the most recent therapy, as defined by one of the following:

   * New soft tissue/visceral/lymph node/bone metastatic lesion
   * Growth of existing soft tissue/visceral/lymph node/bone metastases as determined by the investigator
   * Clinical progression of disease with cutaneous lesions, palpable lesions, pleural effusions, or ascites in absence of radiographic progression
4. Enrollment prior to the initiation of a new systemic therapy.
5. Age > 18 years.
6. Ability to understand and the willingness to sign a written informed consent document.

Colorectal cancer patients will be eligible for inclusion in this study only if all of the following inclusion criteria apply:

1. Histologically confirmed diagnosis of invasive colorectal adenocarcinoma.
2. Clinical or radiographic evidence of metastatic disease.
3. Evidence of disease progression on the current or following the most recent therapy, as defined by one of the following:

   * New soft tissue/visceral/lymph node/bone metastatic lesion
   * Growth of existing soft tissue/visceral/lymph node/bone metastases as determined by the investigator
   * Clinical progression of disease with cutaneous lesions, palpable lesions, pleural effusions, or ascites in absence of radiographic progression
4. Enrollment prior to the initiation of a new systemic therapy.
5. Age > 18 years.
6. Ability to understand and the willingness to sign a written informed consent document.

Pancreatic cancer patients will be eligible for inclusion in this study only if all of the following inclusion criteria apply:

1. Histologically confirmed diagnosis of invasive pancreatic adenocarcinoma.
2. Clinical or radiographic evidence of metastatic disease.
3. Enrollment prior to the initiation of a new systemic therapy.
4. Age > 18 years.
5. Ability to understand and the willingness to sign a written informed consent document.

Advanced, MET amplified, solid tumor patients will be eligible for inclusion in this study only if all of the following inclusion criteria apply:

1. Histologically confirmed diagnosis of cancer (any kind)
2. MET gene amplification by FISH, CISH, rtPCR, or other assay as determined by the investigator.
3. Clinical or radiographic evidence of metastatic disease.
4. Age > 18 years.
5. Ability to understand and the willingness to sign a written informed consent document.

Non-Small Cell Lung Cancer (NSCLC) patients will be eligible for inclusion in this study only if all of the following inclusion criteria apply:

1. Histologically confirmed diagnosis of invasive non-small cell carcinoma of the lung (includes adenocarcinoma, squamous cell carcinoma, large cell carcinoma, adenosquamous, and carcinomas with pleomorphic, sarcomatoid, or sarcomatous elements; does not include carcinoid tumor or neuroendocrine carcinoma).
2. Metastatic disease with either bone or visceral metastatic lesions, or clinically symptomatic with metastatic disease.
3. Progression of disease on or following the most recent treatment as evidenced by one of the following:

   * A new soft tissue/visceral/lymph node/bone metastatic lesion
   * Growth of existing soft tissue/visceral/lymph node/bone metastases as determined by the investigator.
   * Clinical progression of disease with cutaneous lesions or palpable lesions in absence of radiographic progression
4. Progression of disease either on or following treatment with an EGFR inhibitor (such as erlotinib, gefitinib, or other EGFR-targeted therapy)
5. Enrollment prior to the initiation of a new systemic therapy.
6. Age > 18 years.
7. Ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

A patient will not be eligible for inclusion in this study if any of the following criteria apply:

1. History of intercurrent or past medical or psychiatric illness that would make participation in a blood drawing protocol difficult or not feasible at the discretion of the principal investigator or co-investigator(s).
2. Treatment with an anthracycline (including mitoxantrone, doxorubicin, epirubicin, and daunorubicin) within 1 week of CTC collection (applicable in prostate and gastric cancer patients), as anthracyclines cause auto-fluorescence of cells.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2014-03; Primary Completion 2016-05-19 (Actual); Study Completion 2016-07-19 (Actual)

PRIMARY OUTCOMES:
Feasibility | day 1
  Feasibility as measured by successfully detecting at least one CTC in at least 2 out of 10 subjects within each disease site.

SECONDARY OUTCOMES:
Difference in the median number of CTCs | day 1
  The difference in the median number of CTCs detected by each of the capture methods (novel and standard) will be calculated.
Association of the number of detectable CTCs with baseline clinical and pathologic disease characteristics. | day 1
  Within each method, the patient will be used as the unit of observation to describe the association of number of detectable CTC cells with the following baseline characteristics: TNM staging, site of metastases (e.g., bone, liver, lymph nodes), Gleason sum (for PC), PSA (for PC), the number of prior hormone therapies (in PC), CEA (for colorectal cancer), the use of previous EGFR inhibitors and KRAS mutation status (for colorectal cancer), HER2 status and prior HER2 treatments (for gastric cancer), CA 19-9 (for pancreatic cancer), and number of prior chemotherapies.
Kinetics of CTCs over time during treatment with c-MET targeted therapies | 8 weeks
  Change is CTCs in patients with MET amplified tumors undergoing treatment with c-MET targeted therapies will be calculated.

CONTACTS AND LOCATIONS:
Overall Officials: Andrew J Armstrong, MD, Principal Investigator — Duke University
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States